CLINICAL TRIAL: NCT01633372
Title: An Open-Label, Multiple Simon 2-Stage Study of Itacitinib Administered Orally to Subjects With Primary Myelofibrosis (PMF), Post Polycythemia Vera Myelofibrosis (PPV-MF) or Post Essential Thrombocythemia Myelofibrosis (PET-MF)
Brief Title: An Open Label Study of Itacitinib Administered Orally in Patients With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 39110-230
Record Dates: First submitted 2012-06-26; First posted 2012-07-04 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: MPN (Myeloproliferative Neoplasms)
Keywords: Primary Myelofibrosis; PMF; Post Polycythemia Vera Fibrosis; PPV-MF; Post Essential Thrombocythemia Myelofibrosis; PET-MF
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis | interventions — itacitinib; INCB039110

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- itacitinib 100 mg (Experimental): itacitinib 100 mg twice a day
  Interventions: Drug: itacitinib
- itacitinib 200 mg (Experimental): itacitinib 200 mg twice a day
  Interventions: Drug: itacitinib
- itacitinib 300 mg (Experimental): itacitinib 300 mg once a day
  Interventions: Drug: itacitinib
- itacitinib 400 mg (Experimental): itacitinib 400 mg once a day
  Interventions: Drug: itacitinib
- itacitinib 600 mg (Experimental): itacitinib 600 mg once a day
  Interventions: Drug: itacitinib

INTERVENTIONS:
Drug: itacitinib
  Other Names: INCB039110

SUMMARY:
This is a study of itacitinib (INCB039110) in patients with myelofibrosis. This study will evaluate safety and efficacy parameters of itacitinib (INCB039110).

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with PMF, PPV-MF or PET-MF as confirmed by bone marrow biopsy.
* Must score at least 1 point on the Dynamic International Prognostic Scoring System (DIPSS) for prognostic risk factors and have peripheral blast count <10% at both Screening and Baseline hematology assessments.
* Subjects must discontinue all drugs used to treat underlying MF disease no later than Day -14.
* Subjects must have hemoglobin value >/= 8.0g/dL and be willing to receive blood transfusions, have a platelet count >/=50x10^9/L and absolute neutrophil count (ANC) >/= 1x10^9/L.
* Subjects must have palpable spleen or history of splenectomy
* Active symptoms at the screening visit

Exclusion Criteria:

* Women who are pregnant or breastfeeding, and men and women who cannot comply with requirements to avoid fathering a child or becoming pregnant, respectively.
* Subjects with impaired liver function, end stage renal disease on dialysis or clinically significant concurrent infections requiring therapy.
* Subjects with unstable cardiac function or invasive malignancies over the previous 2 years except treated basal or squamous carcinomas of the skin, completely resected intraepithelial carcinoma of the cervix and completely resected papillary thyroid and follicular thyroid cancers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-07-16 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with >/= 50% reduction in total symptom score in each dose group, as measured by the modified The Myelofibrosis Symptom Assessment Form (MFSAF) v3.0 diary | Baseline and Week 12

SECONDARY OUTCOMES:
Proportion of subjects with >/= 35% reduction in spleen volume, and mean percent change in spleen volume | Baseline, Week 12 and Week 24
Proportion of transfusion dependent subjects who exhibit changes in transfusion frequency over any 12 week period on study and proportion of transfusion independent subjects who exhibit changes in hemoglobin level | Baseline to Week 12; Week 13 to Week 24 through the end of study or study termination visit.
Safety and tolerability of itacitinib as measured by adverse events. | Every 4-6 weeks through the end of study or early termination visit (approximately 33 weeks exclusive of the extension phase).

CONTACTS AND LOCATIONS:
Overall Officials: Albert Assad, MD, Study Director — Incyte Corporation
Locations (22):
- United States (14):
  - Birmingham Hematology Oncology Associates, LLC, Birmingham, Alabama
  - Mayo Clinic, Arizona, Scottsdale, Arizona
  - UCLA Hematology & Oncology, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - St Agnes Hospital, Baltimore, Maryland
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Mount Sinai School of Medicine, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - South Carolina Oncology & Associates, Columbia, South Carolina
  - Boston Baskin Cancer Foundation, Inc., Memphis, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Australia (4):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Frankston Hospital, Frankston, Victoria
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
  - St. Mary's Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Mascarenhas JO, Talpaz M, Gupta V, Foltz LM, Savona MR, Paquette R, Turner AR, Coughlin P, Winton E, Burn TC, O'Neill P, Clark J, Hunter D, Assad A, Hoffman R, Verstovsek S. Primary analysis of a phase II open-label trial of INCB039110, a selective JAK1 inhibitor, in patients with myelofibrosis. Haematologica. 2017 Feb;102(2):327-335. doi: 10.3324/haematol.2016.151126. Epub 2016 Oct 27. PMID 27789678